CLINICAL TRIAL: NCT04871217
Title: 68Ga-NODAGA-RGD Cardiac PET in Patients With Acute Myocardial Infarction or Chronic Total Coronary Occlusion
Brief Title: 68Ga-NODAGA-RGD PET in Patients With an Occluded Coronary Artery
Acronym: RGDHeart
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Turku University Hospital (Other Government)
Collaborators: University of Lausanne Hospitals (Other); Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, Antti Saraste, MD, PhD, Turku University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: T02/011/18
Record Dates: First submitted 2021-01-14; First posted 2021-05-04 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Coronary Artery Disease
Keywords: Positron Emission Tomography; Myocardial Infarction
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Acute ST-elevation myocardial infarction or chronic coronary artery occlusion (Experimental): 68-Ga-NODAGA-RGD PET after acute ST-elevation myocardial infarction or before and after re-opening of a chronic coronary artery occlusion
  Interventions: Diagnostic Test: 68Ga-NODAGA-RGD PET-imaging

INTERVENTIONS:
Diagnostic Test: 68Ga-NODAGA-RGD PET-imaging — Patients will undergo cardiac 68Ga-NODAGA-RGD PET in order to detect myocardial αVβ3 integrin expression 3-14 days after an acute myocardial infarction or within 4 weeks before and 2 weeks after re-opening of chronic coronary occlusion. Echocardiography of cardiac function will be performed at the time of PET imaging and repeated 6 months later.

SUMMARY:
Background: In patients with coronary artery disease, acute or chronic coronary artery occlusion is associated with various degrees of ischemic myocardial injury and left ventricle dysfunction. The integrin αVβ3 plays a role in angiogenesis, i.e. formation of new capillaries from pre-existing blood vessels that is increased during repair of ischemic myocardial injury. 68Ga-NODAGA-RGD is a radiopharmaceutical for positron emission tomography (PET) imaging of αVβ3 integrin expression.

Aim: This study aims at evaluating the feasibility of imaging myocardial αVβ3 integrin expression using 68-Ga-NODAGA-RGD PET and whether 68Ga-NODAGA-RGD uptake is associated with myocardial contractile function in patients with an acute or chronic coronary artery occlusion.

Study design: An academic, prospective, open-label study in 60 patients with an acute or chronic coronary occlusion.

Study population: 30 patients with an ST-elevation acute myocardial infarction weeks and left ventricular ejection fraction <50%. 30 patients with planned percutaneous re-opening of a chronic coronary total occlusion and left ventricular ejection fraction <50%.

Study procedures: Patients will undergo cardiac 68Ga-NODAGA-RGD PET within 3 to 14 days after an ST-elevation acute myocardial infarction or within 4 weeks before and 2 weeks after planned percutaneous re-opening of chronic coronary total occlusion. Myocardial perfusion reserve will be evaluated in patients with chronic total occlusion by PET. Echocardiography will be performed at the time of PET imaging and repeated 6 months later to evaluate global and regional left ventricle contractile function. Data on relevant cardiovascular clinical history and blood sample will be obtained at imaging visits. Cardiac events will be evaluated after two years.

End-points: Primary: Myocardial uptake of 68-Ga-NODAGA-RGD after an acute myocardial infarction or before and after opening of chronic coronary occlusion. Secondary: Global and regional left ventricle systolic function. Blood biomarkers of myocardial injury and heart failure. Myocardial perfusion reserve. Adverse cardiac events including death, myocardial infarction, unstable angina pectoris, repeat revascularization and heart failure hospitalizations.

DETAILED DESCRIPTION:
Background: In patients with coronary artery disease, acute or chronic coronary artery occlusion is associated with various degrees of ischemic myocardial injury and left ventricle dysfunction. The integrin αVβ3 plays a role in angiogenesis (Brooks 1994), i.e. formation of new capillaries from pre-existing blood vessels that is increased during repair of ischemic myocardial injury (Meoli 2004, Higuchi 2008, Sherif 2012, Sun 2003, Jenkins 2017). 68Ga-NODAGA-RGD is a radiopharmaceutical for positron emission tomography (PET) imaging of αVβ3 integrin expression (Grönman 2017, Buchegger 2011, Pohle 2012, Gnesin 2017).

Aim: This study aims at evaluating the feasibility of imaging myocardial αVβ3 integrin expression using 68-Ga-NODAGA-RGD PET and whether 68Ga-NODAGA-RGD uptake is associated with myocardial contractile function in patients with an acute or chronic coronary artery occlusion.

Study design: An investigator-initiated, prospective, open-label study in 60 patients with an acute or chronic coronary occlusion.

Study population: 30 patients with an ST-elevation acute myocardial infarction weeks and left ventricular ejection fraction <50%. 30 patients with planned percutaneous re-opening of a chronic coronary total occlusion and left ventricular ejection fraction <50%.

Study procedures: Patients will undergo cardiac 68Ga-NODAGA-RGD PET within 3 to 14 days after an ST-elevation acute myocardial infarction or within 4 weeks before and 2 weeks after planned percutaneous re-opening of chronic coronary total occlusion. Myocardial perfusion reserve will be evaluated in patients with chronic total occlusion by PET myocardial perfusion imaging. Complete echocardiography will be performed at the time of PET imaging and repeated 6 months later to evaluate global and regional left ventricle contractile function. Data on relevant cardiovascular clinical history and blood sample will be obtained at imaging visits. Cardiac events will be evaluated after two years.

Primary end-point: Myocardial uptake of 68-Ga-NODAGA-RGD after an acute myocardial infarction or before and after opening of chronic coronary occlusion. Secondary end-points: Global and regional left ventricle systolic function. Blood biomarkers of myocardial injury (troponin) and heart failure (pro-BNP). Myocardial perfusion reserve. Adverse cardiac events including death, myocardial infarction, unstable angina pectoris, repeat revascularization and heart failure hospitalizations.

Sample size: This is an exploratory study and formal power calculation cannot be performed.

Ethical aspects: The study conforms to the World Medical Association Declaration of Helsinki. Written statement will be obtained from the ethics committee (the Ethical Board of the South-Western Finland). Permissions from regulatory authorities (the Finnish Medicines Agency Fimea) and the Turku University Hospital for conducting the study will be obtained. Signed and dated informed consent will be obtained from patients before conducting any study specific procedures.

ELIGIBILITY:
Inclusion Criteria:

* ST-elevation acute myocardial infarction within 3-14 days
* Planned elective percutaneous revascularization of angiographically documented coronary chronic total occlusion (CTO)
* Left ventricular ejection fraction < 50% when hospitalized for index acute myocardial infarction or within 12 months before planned revascularization of coronary CTO
* Provision of signed and dated informed consent prior to study specific procedures

Exclusion Criteria:

* Current unstable angina
* Significant valvular heart disease
* NYHA IV heart failure symptoms
* Severe untreated hypertension (>180/110 mmHg)
* Female not post-menopausal
* Contraindications for adenosine infusion (in patients with CTO):
* Severe renal failure (estimated glomerular filtration rate < 30 ml/min)
* Atrial fibrillation with ventricular response > 110 bpm
* No acoustic window for left ventricle assessment by echocardiography
* Previous cardiac surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-12-04 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Myocardial uptake of 68Ga-NODAGA-RGD after acute myocardial infarction | 3 to 14 days after acute myocardial infarction
  68Ga-NODAGA-RGD uptake in PET images in the myocardial territory supplied by the occluded coronary artery vs. remote myocardium after an acute myocardial infarction
Myocardial uptake of 68Ga-NODAGA-RGD before and after opening of chronic coronary occlusion | Within 4 weeks before and 2 weeks after re-opening of a chronic coronary occlusion
  Change in 68Ga-NODAGA-RGD uptake in PET images in the myocardial territory supplied by the occluded coronary artery before and after opening of a chronic coronary occlusion

SECONDARY OUTCOMES:
Global left ventricle systolic function | At the time of 68Ga-NODAGA-RGD PET imaging and after 6 months of follow-up
  Left ventricle ejection fraction (%) assessed by echocardiography
Regional left ventricle systolic function | At the time of 68Ga-NODAGA-RGD PET imaging and after 6 months of follow-up
  Regional myocardial strain (%) assessed by echocardiography
Myocardial perfusion reserve | At the time of 68Ga-NODAGA-RGD PET imaging within 4 weeks before and 2 weeks after re-opening of a chronic coronary occlusion
  Assessed by PET myocardial perfusion imaging before and after re-opening of chronic coronary occlusion
Adverse cardiac events | After 2 years of follow-up
  Number of patients with myocardial infarction, unstable angina pectoris, repeat revascularization, heart failure hospitalization or death
Blood biomarker of heart failure | At the time of 68Ga-NODAGA-RGD PET imaging and after 6 months of follow-up
  pro-BNP (ng/L)
Blood biomarker of myocardial injury | At the time of 68Ga-NODAGA-RGD PET imaging and after 6 months of follow-up
  Cardiac troponin T (ng/L)

CONTACTS AND LOCATIONS:
Overall Officials: Antti Saraste, MD, PhD, Principal Investigator — Turku University Hospital
Locations (3):
- Turku University Hospital, Turku, Finland
- Leiden Medical Center, Leiden, Netherlands
- University of Lausanne Hospitals, Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: No
May be shared upon reasonable request to the PI

REFERENCES:
- [Background] Brooks PC, Clark RA, Cheresh DA. Requirement of vascular integrin alpha v beta 3 for angiogenesis. Science. 1994 Apr 22;264(5158):569-71. doi: 10.1126/science.7512751.
- [Background] Buchegger F, Viertl D, Baechler S, Dunet V, Kosinski M, Poitry-Yamate C, Ruegg C, Prior JO. 68Ga-NODAGA-RGDyK for alphavbeta3 integrin PET imaging. Preclinical investigation and dosimetry. Nuklearmedizin. 2011;50(6):225-33. doi: 10.3413/Nukmed-0416-11-06. Epub 2011 Oct 11. PMID 21989840
- [Background] Gronman M, Tarkia M, Kiviniemi T, Halonen P, Kuivanen A, Savunen T, Tolvanen T, Teuho J, Kakela M, Metsala O, Pietila M, Saukko P, Yla-Herttuala S, Knuuti J, Roivainen A, Saraste A. Imaging of alphavbeta3 integrin expression in experimental myocardial ischemia with [68Ga]NODAGA-RGD positron emission tomography. J Transl Med. 2017 Jun 19;15(1):144. doi: 10.1186/s12967-017-1245-1. PMID 28629432
- [Background] Higuchi T, Bengel FM, Seidl S, Watzlowik P, Kessler H, Hegenloh R, Reder S, Nekolla SG, Wester HJ, Schwaiger M. Assessment of alphavbeta3 integrin expression after myocardial infarction by positron emission tomography. Cardiovasc Res. 2008 May 1;78(2):395-403. doi: 10.1093/cvr/cvn033. Epub 2008 Feb 6. PMID 18256073
- [Background] Jenkins WS, Vesey AT, Stirrat C, Connell M, Lucatelli C, Neale A, Moles C, Vickers A, Fletcher A, Pawade T, Wilson I, Rudd JH, van Beek EJ, Mirsadraee S, Dweck MR, Newby DE. Cardiac alphaVbeta3 integrin expression following acute myocardial infarction in humans. Heart. 2017 Apr;103(8):607-615. doi: 10.1136/heartjnl-2016-310115. Epub 2016 Dec 7. PMID 27927700
- [Background] Meoli DF, Sadeghi MM, Krassilnikova S, Bourke BN, Giordano FJ, Dione DP, Su H, Edwards DS, Liu S, Harris TD, Madri JA, Zaret BL, Sinusas AJ. Noninvasive imaging of myocardial angiogenesis following experimental myocardial infarction. J Clin Invest. 2004 Jun;113(12):1684-91. doi: 10.1172/JCI20352. PMID 15199403
- [Background] Pohle K, Notni J, Bussemer J, Kessler H, Schwaiger M, Beer AJ. 68Ga-NODAGA-RGD is a suitable substitute for (18)F-Galacto-RGD and can be produced with high specific activity in a cGMP/GRP compliant automated process. Nucl Med Biol. 2012 Aug;39(6):777-84. doi: 10.1016/j.nucmedbio.2012.02.006. Epub 2012 Mar 22. PMID 22444238
- [Background] Sherif HM, Saraste A, Nekolla SG, Weidl E, Reder S, Tapfer A, Rudelius M, Higuchi T, Botnar RM, Wester HJ, Schwaiger M. Molecular imaging of early alphavbeta3 integrin expression predicts long-term left-ventricle remodeling after myocardial infarction in rats. J Nucl Med. 2012 Feb;53(2):318-23. doi: 10.2967/jnumed.111.091652. PMID 22302965
- [Background] Sun M, Opavsky MA, Stewart DJ, Rabinovitch M, Dawood F, Wen WH, Liu PP. Temporal response and localization of integrins beta1 and beta3 in the heart after myocardial infarction: regulation by cytokines. Circulation. 2003 Feb 25;107(7):1046-52. doi: 10.1161/01.cir.0000051363.86009.3c. PMID 12600920
- [Background] Gnesin S, Mitsakis P, Cicone F, Deshayes E, Dunet V, Gallino AF, Kosinski M, Baechler S, Buchegger F, Viertl D, Prior JO. First in-human radiation dosimetry of 68Ga-NODAGA-RGDyK. EJNMMI Res. 2017 Dec;7(1):43. doi: 10.1186/s13550-017-0288-x. Epub 2017 May 18. PMID 28523582
- [Derived] Nammas W, Paunonen C, Teuho J, Siekkinen R, Luoto P, Kakela M, Hietanen A, Viljanen T, Dietz M, Prior JO, Li XG, Roivainen A, Knuuti J, Saraste A. Imaging of Myocardial alphavbeta3 Integrin Expression for Evaluation of Myocardial Injury After Acute Myocardial Infarction. J Nucl Med. 2024 Jan 2;65(1):132-138. doi: 10.2967/jnumed.123.266148. PMID 37973184